CLINICAL TRIAL: NCT06308276
Title: Effects of Aerobic Versus Resistance Training on Blood Pressure, Cardiorespiratory Fitness and Quality of Life in Post Percutaneous Coronary Intervention Obese Patients
Brief Title: Effects of Aerobic Versus Resistance Training in Post Percutaneous Coronary Intervention Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0363
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases
Keywords: Aerobic Exercise; Angioplasty; Obese Patients; Percutaneous Coronary Intervention; Resistance Training
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Brisk walking, jogging, cycling, or low-impact aerobics
  Interventions: Other: Aerobic Training
- Group B (Active Comparator): Full body resistance exercise targeting major muscle groups, including squats, lunges, chest presses, rows, and core exercises
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Aerobic Training — Aerobic Training: Brisk walking, jogging, cycling, or low-impact aerobics
  Arms: Group A
Other: Resistance Training — Resistance Training: Full body resistance exercise targeting major muscle groups, including squats, lunges, chest presses, rows, and core exercises
  Arms: Group B

SUMMARY:
The randomized clinical trial (RCT) endeavors to enroll 50 participants, divided equally into aerobic exercise and resistance exercise groups. The study employs rigorous tools such as blood pressure measurement, SF-36 questionnaire, and the Six-Minute Walk Test (6MWT) to assess VO2max.

DETAILED DESCRIPTION:
The randomized clinical trial (RCT) endeavors to enroll 50 participants, divided equally into aerobic exercise and resistance exercise groups. The non-probability convenient sampling technique, followed by random allocation using a lottery method, ensures a diverse yet unbiased sample. Will be conducted at the Sialkot Medical and Physiotherapy Centre, the inclusion criteria will focus on post-PCI patients aged 40-60, presenting with a BMI of 30 or higher. The study employs rigorous tools such as blood pressure measurement, SF-36 questionnaire, and the Six-Minute Walk Test (6MWT) to assess VO2max. The aerobic exercise group undergoes sessions three times a week, progressively increasing in duration and intensity, emphasizing activities like brisk walking and cycling. The resistance exercise group follows a similar schedule, engaging in full-body resistance exercises targeting major muscle groups. Both groups undergo assessments using cardiopulmonary exercise testing (CPET) to determine exercise tolerance accurately.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 40 and 60 years old.
* Gender: Male and female both.
* Cardiovascular Status: Post Percutaneous Coronary Intervention (PCI) patients with a documented history of coronary artery disease
* Participants who are at least three months post PCI to ensure stabilization of their cardiovascular condition.
* Obesity: Participants must have a Body Mass Index (BMI) equal to or greater than 30 kg/m², indicating obesity.
* Health Status: Participants should be in stable health condition to participate in moderate physical activities.
* Willingness to Participate: Participants must provide informed consent and be willing to comply with the study protocol, including attending scheduled exercise sessions and follow-up assessments.
* Participants capable of engaging in either aerobic or resistance training, were assessed by a physical activity readiness questionnaire (PAR-Q).

Exclusion Criteria:

* Participants with severe physical limitations, disabilities, or musculoskeletal disorders that would prevent them from engaging in aerobic and resistance exercises.
* Individuals with a history of substance abuse or current substance abuse issues that might interfere with their ability to participate or adhere to the study protocol.
* Patients with Neurological diseases
* Patients with severe or unstable heart conditions, recent heart attack, or heart failure

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 4 Weeks
  Blood pressure is a crucial physiological parameter often employed as a data collection tool in research, particularly in studies focused on cardiovascular health and related interventions.
Six Minute Walk Test | 4 Weeks
  The 6-minute walk test (6MWT) serves as a valuable and widely used data collection tool in research, particularly in studies assessing functional capacity, exercise tolerance, and overall physical performance.
SF 36 Questionnaire | 4 Weeks
  The Short Form 36 (SF-36) is a widely used health-related quality of life (HRQoL) questionnaire that serves as a comprehensive data collection tool in research studies across various disciplines.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faizan Hamid, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Sialkot Medical and Physiotherapy Center, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No